CLINICAL TRIAL: NCT01829061
Title: Reproducibility and Method Comparison of the Quo-Test™ A1C System and the Quo-Lab A1C Test and CLIA Waiver of the Quo-Test™ A1C System
Brief Title: Reproducibility and Method Comparison Studies of the Quo-Test™ A1C System and the Quo-Lab A1C Test and CLIA Waiver Study of the Quo-Test™ A1C System
Status: Terminated | Type: Observational
Why Stopped: Data for Study Devices vs. Predicate not within allowable ranges.
Sponsor: Quotient Diagnostics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: QDL Clinical Studies
Record Dates: First submitted 2013-04-01; First posted 2013-04-11 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes
Keywords: Type I Diabetes; Type II Diabetes; HbA1C
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Whole Blood Venous Draw and Capillary Blood - IVD Study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment

SUMMARY:
The Quo-Test A1C Analyzer and Reagent Test System (Quo-Test A1C System) are intended for the in-vitro quantitative determination of glycated hemoglobin in whole blood samples obtained from fingerstick or venous samples for point-of-care testing. The Quo-Test A1C System is indicated in the management and treatment of diabetes and for monitoring long term glycemic control by diabetics. It is for multiple patient use. Only auto-disabling, single use lancing devices should be used with this system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Able to read English
* Read, understood and signed the Informed Consent Form
* Agrees to participate and does not withdraw\
* Either healthy (without diabetes) or has Type 1 or Type 2 diabetes

Exlcusion Criteria:

• Declines participation or withdraws before study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From site's patient database
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The objective is to conduct reproducibility testing using duplicates of each of 3 levels of HbA1C | 10 Days
  The objective is to conduct a method comparison between both the Quo-Test and Quo-Lab investigational devices and the reference method [Tosoh G8 (K071132)]. The reference method also serves as the predicate for the premarket notifications for both investigational devices. Both capillary and venous samples will be tested on the Quo-Test A1C System and Quo-Lab A1C Test, while only venous samples will be tested on the reference method.

SECONDARY OUTCOMES:
Obtain CLIA Waiver Status for the Quo-Test | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bailey, MD, Principal Investigator — AMCR Institute; Stephanie Svoboda, PharmD, Principal Investigator — Ridgeview Research; Michael Gardner, MD, Principal Investigator — University of Missouri-Columbia
Locations (3):
- United States (3):
  - AMCR Institute, Escondido, California
  - Ridgeview Research, Chaska, Minnesota
  - University of Missouri, Columbia, Missouri